CLINICAL TRIAL: NCT03069833
Title: Computer Aided Diagnosis of Colorectal Neoplasms During Colonoscopic Examination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Peng-Jen Chen, Head of Endoscopy Center, Tri-Service General Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2-105-05-061
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Colon Polyp
MeSH Terms: conditions — Colonic Polyps | interventions — Diagnosis, Computer-Assisted

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer-aided diagnosis (Experimental)
  Interventions: Diagnostic Test: Computer-aided diagnosis
- traditional diagnosis (No Intervention)

INTERVENTIONS:
Diagnostic Test: Computer-aided diagnosis — computer-aided diagnosis to assist colonoscopists
  Arms: Computer-aided diagnosis

SUMMARY:
An NBI-based diagnosis requires training and experience. We are developing a system of computerized image recognition, which can detect possible NBI features of polyps, and provide a more objective diagnosis, which allows nonexpert endoscopists to achieve a high diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

the same as colonoscopy

Exclusion Criteria:

the same as colonoscopy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, Specificity, False Positive, False Negative | Duration between endoscopic diagnosis and pathologic diagnosis is about one week
  Diagnostic accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Peng-Jen Chen, MD, Principal Investigator — Tri-Service General Hospital, National Defense Medical Center, Taiwan
Locations (1):
- Endoscopy Center, Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided